CLINICAL TRIAL: NCT07018375
Title: The Effect of Oliceridine Patient-Controlled Intravenous Analgesia on Postoperative Chronic Pain After Video-Assisted Thoracoscopic Lobectomy
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Tianjin Medical University General Hospital (Other)
Responsible Party: Principal Investigator, Yang Jiao, Associate Chief Physician, Tianjin Medical University General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB2025-YX-199-01
Record Dates: First submitted 2025-05-27; First posted 2025-06-12 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Chronic Postsurgical Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — ((3-methoxythiophen-2-yl)methyl)((2-(9-(pyridin-2-yl)-6-oxaspiro(4.5)decan-9-yl)ethyl))amine; Sufentanil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oliceridine group (Experimental): Administer a loading dose of 0.03 mg/kg intravenously 20-30 minutes before the end of surgery. Postoperative PCA pump configuration: 0.6 mg/kg oxycodone diluted with normal saline to a total volume of 100 mL, with a background infusion rate of 2 mL/h, PCA bolus dose of 0.5 mL per injection, lockout interval of 15 minutes, and treatment duration of 48 hours.
  Interventions: Drug: Oliceridine
- Sufentanil Group (Active Comparator): Administer a loading dose of 0.1 μg/kg intravenously 20-30 minutes before the end of surgery. Postoperative PCA pump configuration: 2 μg/kg sufentanil diluted with normal saline to a total volume of 100 mL, with a background infusion rate of 2 mL/h, PCA bolus dose of 0.5 mL per injection, lockout interval of 15 minutes, and treatment duration of 48 hours.
  Interventions: Drug: Sufentanil

INTERVENTIONS:
Drug: Oliceridine — postoperative patient-controlled analgesia (PCA)
  Arms: Oliceridine group
Drug: Sufentanil — Sufentanil
  Arms: Sufentanil Group

SUMMARY:
The primary objective is to evaluate the impact of oliceridine versus sufentanil for perioperative analgesia on the incidence of chronic postsurgical pain (CPSP) in patients undergoing video-assisted thoracoscopic surgery.

DETAILED DESCRIPTION:
The primary objective is to evaluate the impact of oliceridine administered via patient controlled analgesia device（PCA）versus sufentanil administered via PCA on the incidence of chronic postsurgical pain (CPSP) in patients undergoing video-assisted thoracoscopic surgery.

ELIGIBILITY:
Inclusion Criteria:

* ① Age 18-75 years, ASA physical status I-III, BMI 18-30 kg/m²;

  * Scheduled for unilateral video-assisted thoracoscopic surgery (VATS) lung resection, including wedge resection, segmentectomy, lobectomy, or radical resection for lung cancer;

    * Preoperative pain score <1 on the Numeric Rating Scale (NRS);

      * Ability to understand the study objectives and procedures, with voluntary informed consent obtained;

        * Expected postoperative recovery in the general ward setting.

Exclusion Criteria:

* ① History of chronic pain or long-term analgesic use prior to surgery;

  * Previous ipsilateral thoracic surgery;

    * Prior neoadjuvant radiotherapy or chemotherapy;

      * Severe cardiovascular or cerebrovascular disease, or hepatic/renal dysfunction (ALT/AST >3× upper limit of normal; eGFR <60 mL/min/1.73m²);

        * Concurrent malignancy or active infection;

          * Pre-existing psychiatric disorders or communication barriers precluding study participation;

            * Known hypersensitivity to study medications (opioids, adjuvant analgesics, anesthetics, or antiemetics);

              * Any condition deemed unsuitable for study participation by the investigator

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2026-01-06 (Estimated); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of chronic pain after surgery | from day 1 to day 90 after surgery
  Chronic pain intensity was assessed by a numeric rating scale (NRS) using a telephone questionnaire

SECONDARY OUTCOMES:
postoperative acute pain NRS scoring | 24h and 48h after surgery
  Acute pain NRS score (rest versus cough) at 24 and 48 hours after surgery
Incidence of adverse events | 48 hours after surgery
Chronic pain NRS score 3 months after surgery | 3 months postoperatively
  assessed by NRS scale
Neuropathic pain (DN4 score ≥ 4) | 1 day preoperatively；3 months postoperatively
  the DN4 questionnaire is a brief and user-friendly screening tool designed to identify the presence of neuropathic pain components
Sleep quality assessment | 1 day preoperatively；3 months postoperatively
  By Pittsburgh Sleep Index (PSQI) scale
Psychological status assessment | 1 day preoperatively； 3 months postoperatively
  By Hamilton Anxiety/Depression Rating Scale (HAMA/HADS)
Evaluate pain catastrophizing levels in surgical patients | 1 day preoperatively；3 months postoperatively
  By PCS Scale
Quality of Life Assessments | 1 day preoperatively；3 months postoperatively
  The 36-Item Short Form Survey (SF-36)
Use and frequency of rescue analgesic administration | 1 day preoperatively；3 months postoperatively
  Dose and frequency of rescue analgesics

CONTACTS AND LOCATIONS:
Overall Officials: Yang Jiao, Doctor, Principal Investigator — Tianjin Medical University General Hospital

IPD SHARING:
Plan to Share IPD: No